CLINICAL TRIAL: NCT04385420
Title: Phase 1 Single Dose Escalation/Multiple Dose Escalation Study to Evaluate the Safety, Tolerability, And Pharmacokinetics of Ascending Doses of a MEK Inhibitor (ATR-002) Given for 7 Days in Healthy Subjects
Brief Title: Phase 1 Study of ATR-002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atriva Therapeutics GmbH (Industry)
Collaborators: SGS Life Sciences, a division of SGS Belgium NV (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATR002-01
Record Dates: First submitted 2020-05-06; First posted 2020-05-12 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: This was a combination of a single ascending dose (SAD) study to evaluate the safety, tolerability, and PK of 3 oral doses of a MEK inhibitor and a multiple ascending dose (MAD) study of 3 oral doses of a MEK inhibitor.
  Subjects were to be enrolled in 3 different cohorts in the SAD and 3 different cohorts in the MAD and were to be randomly (blinded) allocated to active treatment or placebo (each cohort consisted of 8 subjects receiving active treatment and 2 subjects receiving placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Between each cohort, a blinded interim analysis of PK, safety and tolerability had to be performed. The available data was evaluated by the Investigator and sponsor in a Safety Review Committee (SRC) meeting.
  Once a dose level was judged to be safe, the SRC determined the dose level for the next cohort considering a maximal increment of 400 mg compared to the previous cohort, and the next dose level could be administered to the next cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- ATR-002 100 mg (SAD) (Experimental): 100 mg ATR-002 once (morning)
  Interventions: Drug: ATR-002 MEK Inhibitor
- ATR-002 300 mg (SAD) (Experimental): 300 mg ATR-002 once (morning)
  Interventions: Drug: ATR-002 MEK Inhibitor
- ATR-002 600 mg (SAD) (Experimental): 600 mg ATR-002 once (morning)
  Interventions: Drug: ATR-002 MEK Inhibitor
- ATR-002 900 mg (SAD) (Experimental): 900 mg ATR-002 once (morning)
  Interventions: Drug: ATR-002 MEK Inhibitor
- Placebo (SAD) (Placebo Comparator): Placebo once (morning)
  Interventions: Drug: Placebo oral tablet
- ATR-002 100 mg (MAD) (Experimental): 100 mg ATR-002 once daily (morning) for 7 days
  Interventions: Drug: ATR-002 MEK Inhibitor
- ATR-002 300 mg (MAD) (Experimental): 300 mg ATR-002 once daily (morning) for 7 days
  Interventions: Drug: ATR-002 MEK Inhibitor
- ATR-002 600 mg (MAD) (Experimental): 600 mg ATR-002 once daily (morning) for 7 days
  Interventions: Drug: ATR-002 MEK Inhibitor
- Placebo (MAD) (Placebo Comparator): Placebo once daily (morning) for 7 days
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: ATR-002 MEK Inhibitor — Drug ATR-002 administered as film-coated tablet via oral route
  Other Names: PD01842649
  Arms: ATR-002 100 mg (MAD); ATR-002 100 mg (SAD); ATR-002 300 mg (MAD); ATR-002 300 mg (SAD); ATR-002 600 mg (MAD); ATR-002 600 mg (SAD); ATR-002 900 mg (SAD)
Drug: Placebo oral tablet — Placebo film-coated tablet administered via oral route
  Arms: Placebo (MAD); Placebo (SAD)

SUMMARY:
This was a combination of a single ascending dose (SAD) study to evaluate the safety, tolerability, and PK of 3 oral doses of a MEK inhibitor and a multiple ascending dose (MAD) study of 3 oral doses of a MEK inhibitor.

Subjects were to be enrolled in 3 different cohorts in the SAD and 3 different cohorts in the MAD and were to be randomly (blinded) allocated to active treatment or placebo (each cohort consisted of 8 subjects receiving active treatment and 2 subjects receiving placebo).

DETAILED DESCRIPTION:
Each subject in the SAD cohorts was to receive a single dose of the MEK inhibitor ATR-002 (PD0184264), with a starting dose of 100 mg ATR-002 or placebo:

* Cohort 1: 100 mg ATR-002 or placebo;
* Cohort 2: 100 mg + X mg ATR-002 or placebo;
* Cohort 3: 100 mg + X mg + Y mg ATR-002 or placebo. An additional cohort (Cohort 4) of 10 subjects (4:1 active vs placebo) could have been recruited into the SAD Part, if appropriate.

Effectively, 4 cohorts were treated:

* Cohort 1: 100 mg ATR-002 or placebo;
* Cohort 2: 300 mg ATR-002 or placebo;
* Cohort 3: 600 mg ATR-002 or placebo;
* Cohort 4: 900 mg ATR-002 or placebo. Between each cohort, a blinded interim analysis of PK, safety and tolerability had to be performed. The available data was evaluated by the Investigator and sponsor in a Safety Review Committee (SRC) meeting.

Once a dose level was judged to be safe, the SRC determined the dose level for the next cohort considering a maximal increment of 400 mg compared to the previous cohort, and the next dose level could be administered to the next cohort.

The maximal dose level could not exceed 900 mg ATR-002. Each subject in the MAD cohorts was to receive once daily (QD) doses (fasted) of the MEK inhibitor ATR-002 for 7 days, starting with a dose of 100 mg ATR-002 or placebo QD.

* Cohort 5: 100 mg ATR-002 QD or placebo;
* Cohort 6: 100 mg + A mg ATR-002 QD or placebo;
* Cohort 7: 100 mg + A mg + B mg ATR-002 QD or placebo. An additional cohort (Cohort 8) of 10 subjects (4:1 active vs placebo) could be recruited into the MAD Part, if appropriate.

Effectively, 3 cohorts were treated:

* Cohort 5: 100 mg ATR-002 QD or placebo;
* Cohort 6: 300 mg ATR-002 QD or placebo;
* Cohort 7: 600 mg ATR-002 QD or placebo. Between each cohort, a blinded interim analysis of PK, safety and tolerability had to be performed. The available data was evaluated by the Investigator and sponsor in a SRC meeting. Once a dose level was judged to be safe, the SCR determined the dose level for the next cohort considering a maximal increment of 400 mg compared to the previous cohort, and the next dose level could be administered to the next cohort.

The maximal dose level could not exceed 900 mg ATR-002. During the study, no repeated daily dose could exceed the maximum single dose that has been shown to cause no safety concerns.

Subjects were resident on the ward from the day (late afternoon/evening) before dosing (Day -1) until completion of procedures at 96h following their final dose of study medication. They were to attend a follow up visit 28 days (± 2 days) following their final dose of study medication.

Subjects with AEs that were ongoing at the end of the study were followed up as appropriate until the AEs had resolved or stabilised, up to a maximum of 30 days after the last dose of study drug.

Pharmacokinetics were determined predose 30 min, 1h, 2h, 4h, 8h, 12h, and 24h, postdose, and predose on Day 2-4 in the SAD Part, and predose 30 min, 1h, 2h, 4h, 8h, 12h, and 24h, of Day 1 and Day 7, predose on Day 2-6 and 48h, 72h, and 96h post final dose of Day 7 in the MAD Part. The 72h and 96h samples in both SAD and MAD were only to be analysed if deemed informative based on the results of the 48h PK sample.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, between 18 and 55 years old, extremes included;
2. Weighed at least 50 kg and had a body mass index (BMI) within normal range: 18.0≤ BMI <31.0 kg/m2;
3. In good physical and mental health as determined on the basis of medical history and general physical examination performed at screening;
4. Haematology and chemistry parameters, pulse rate and/or blood pressure, and ECG within the reference range for the population studied, or showing no clinically relevant deviations, as judged by the Investigator;
5. Negative urine test for selected drugs of abuse at screening and upon check-in at the clinical site; Note: Subjects could not consume poppy-seeds within 24h before screening and before each urine drug screening because this could falsify the results of the opiate urine drug test.
6. Negative alcohol breath test at screening and upon check-in at the clinical site;
7. Negative hepatitis panel (including hepatitis B surface antigen [HBsAg] and anti hepatitis C virus [HCV] antibodies) and negative human immunodeficiency virus (HIV) antibody screens;
8. Female subjects had to be of non-childbearing potential, as follows:

   1. At least 1 year post-menopausal (amenorrhea >12 months in the absence of an alternative medical cause and follicle-stimulating hormone >30 mIU/mL in women not using hormonal contraception or hormonal replacement therapy) prior to screening;
   2. Surgically sterile (bilateral oophorectomy, hysterectomy, bilateral salpingectomy, or bilateral tubal ligation);
9. To protect partners from possible exposure to study medication in semen, male subjects had to use a condom during the study, even if they had a vasectomy or their partner was not of childbearing potential.

   Note: medically acceptable methods of contraception that could be used by the partner included combined oral contraceptive, contraceptive vaginal ring, contraceptive injection, intrauterine device, and etonogestrel implant;
10. Willing to adhere to the prohibitions and restrictions specified in the protocol (see Appendix 16.1.1);
11. Ability to comprehend the nature of the study and any hazards of participating in it. Ability to communicate satisfactorily with the Investigator and to participate in, and comply with the requirements of, the entire study;
12. Informed Consent Form (ICF) signed voluntarily before any study-related procedure was performed, indicating that the subject understood the purpose of and procedures required for the study and was willing to participate in the study.

Exclusion Criteria:

1. Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-study screening assessment that could interfere with the objectives of the study or the safety of the subject;
2. Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the subject's participation in the study or make it unnecessarily hazardous;
3. A condition that, in the opinion of the Investigator, could compromise the well being of the subject or course of the study, or prevent the subject from meeting or performing any study requirements;
4. Impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease, cancer, or history of any psychotic mental illness;
5. Respiratory tract infection within 4 weeks before the screening visit;
6. History of surgery or medical intervention, or planned surgery or medical intervention, that could interfere with the objectives of the study or the safety of the subject;
7. Presence or history of severe adverse reaction to any drug, or sensitivity to components of the study medication;
8. Use of a prescription or over-the-counter medicine, with the exception of acetaminophen (paracetamol), during the 7 days (or 5 half-lives, whichever is longer) before the first dose of study medication;
9. Participation in another clinical study of a new chemical entity, new device, or a prescription medicine within the 3 months before dosing, or participation within 5 half-lives of receiving an experimental drug (whichever is longer);
10. Presence or history of drug or alcohol abuse, or intake of more than 21 units (14 units for women) of alcohol weekly;
11. Use of a prohibited therapy;
12. Current smoker; or ex-smokers who (a) gave up less than 1 year ago, or (b) who had a history of more than 10 pack-years; Pack-years = cigarettes per day x number of years smoked/20
13. Blood pressure and heart rate at the screening examination outside the ranges 90 150 mmHg systolic, 40-90 mmHg diastolic; heart rate 40-100 bpm;
14. Loss of more than 400 mL blood, e.g. as a blood donor, or donation of blood products, during the 3 months before the study;
15. History of tuberculosis infection;
16. Receipt of a living vaccine within the 3 months before dosing;
17. Active or latent parasitic infection, visit to a country with a high prevalence of parasitic infections within 3 months before receiving study medication;
18. Positive faecal blood test at screening;
19. Employee of the Investigator or the Sponsor, who was directly involved in the study, or a first-degree relative of such person;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAE) - SAD | Day 1- Day 5
  TEAEs in SAD groups
Treatment-emergent adverse events (TEAE) - MAD | Day 1 - Day 11
  TEAEs in MAD groups

SECONDARY OUTCOMES:
Maximum plasma concentration - Cmax (SAD) | Day 1- Day 5
  Cmax in SAD groups
Time to maximum plasma concentration tmax (SAD) | Day 1- Day 5
  Tmax in SAD groups
Area under plasma concentration AUC0-t (SAD) | Day 1- Day 5
  AUC0-t in SAD groups
Area under plasma concentration AUC0-inf (SAD) | Day 1- Day 5
  AUC0-inf in SAD groups
Elimination half-life t1/2 (SAD) | Day 1- Day 5
  t1/2 in SAD groups
Maximum plasma concentration - Cmax (MAD) | Day 1 - Day 11
  Cmax in MAD groups
Time to maximum plasma concentration tmax (MAD) | Day 1 - Day 11
  Tmax in MAD groups
Area under plasma concentration AUC0-t (MAD) | Day 1 - Day 11
  AUC0-t in MAD groups
Area under plasma concentration AUC0-tau (MAD) | Day 1 - Day 11
  AUC0-tau in MAD groups
Minimum plasma concentration Ctrough (MAD) | Day 1 - Day 11
  Ctrough in MAD groups
Area under plasma concentration AUC0-inf (MAD) | Day 1 - Day 11
  AUC0-inf in MAD groups
Elimination half-life t1/2 (MAD) | Day 1 - Day 11
  T1/2 in MAD groups
Accumulation ratio Cmax (MAD) | Day 1 - Day 11
  Cmax Accumulation in MAD groups
Accumulation ratio AUC0-tau (MAD) | Day 1 - Day 11
  AUC0-tau accumulation ratio in MAD groups
Accumulation ratio Ctrough (MAD) | Day 1 - Day 11
  Ctrough accumulation ratio in MAD groups

CONTACTS AND LOCATIONS:
Overall Officials: Bram Volckaert, MD, Principal Investigator — SGS Belgium NV
Locations (1):
- SGS Life Sciences, Clinical Pharmacology Unit Antwerpen, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No